CLINICAL TRIAL: NCT00778726
Title: Single Dose Two-Way Crossover Fasted Bioequivalence Study of Benazepril HCl/ Hydrochlorothiazide 20 mg/ 25 mg Tablets in Healthy Volunteers
Brief Title: Bioequivalence Study of Benazepril HCl / Hydrochlorothiazide 20 mg/ 25 mg Tablets Under Fasting Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research labs
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AAI-US-256
Record Dates: First submitted 2008-10-22; First posted 2008-10-23 (Estimated); Last update posted 2008-10-23 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: Bioequivalence benazepril and hydrochlorothiazide tablets
MeSH Terms: interventions — benazepril; Hydrochlorothiazide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Benazepril HCl/ Hydrochlorothiazide 20 mg/ 25 mg Tablets of Ranbaxy
  Interventions: Drug: Benazepril HCl/ Hydrochlorothiazide 20 mg/ 25 mg Tablets
- 2 (Active Comparator): Lotensin® HCT tablets
  Interventions: Drug: Benazepril HCl/ Hydrochlorothiazide 20 mg/ 25 mg Tablets

INTERVENTIONS:
Drug: Benazepril HCl/ Hydrochlorothiazide 20 mg/ 25 mg Tablets

SUMMARY:
The purpose of this study was to determine the bioavailability of benazepril and hydrochlorothiazide (HCTZ) from two Benazepril/HCTZ 20 mg/25 mg products after administration of single doses to normal healthy fasted subjects. These data were to be evaluated statistically to determine if the products meet bioequivalence criteria.

DETAILED DESCRIPTION:
The study was performed as a single-dose (one 20 mg/25 mg tablet), two way crossover bioequivalence study with a wash out of 7 days between doses and with equal number of subjects randomly assigned to the sequence (AB or BA) in which they received the study Test (A) and Reference (B) treatments.

Subjects were confined in the clinical facility for at least 10 hours before dosing and for 24 hours after dosing. Subjects were discharged after 24-hours blood sample and returned as outpatients for the remaining blood samples. Standardized meals were served and no caffeine, alcohol, or grapefruit-containing foods or beverages were allowed to be consumed 24 hours before dosing or throughout study confinement.

A total of 42 non-smoking subjects (24 men and 18 women) were randomized to receive single oral dose of Benazepril HCl/ Hydrochlorothiazide 20 mg/ 25 mg tablet and 41 subjects completed both the periods of the study.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Subjects at least 18 years of age.
* Informed of the nature of the study and given written informed consent.
* Have a body weight within 15% of the appropriate range as defined in the 1983 Metropolitan Life Company tables weighing at least 110 pounds.

Exclusion Criteria:

* - Hypersensitivity to benazepril (Lotensin®) or thiazide diuretics such as hydrochlorothiazide (Oretic®).
* Any history of clinical condition that might affect drug absorption, metabolism or excretion.
* Recent history (within one year) of mental illness, drug addiction, drug abuse or alcoholism.
* Donation of greater than 500 ml of blood in the past 4 weeks prior to study dosing or difficulty in donating blood.
* Received an investigational drug within the past 4 weeks prior to study dosing.
* Currently taking any prescription medication, except for oral contraceptives, within the 7 days prior to study dosing or over -the counter medication within 3 days of study dosing. This prohibition does not include vitamins or herbal preparations taken as nutritional supplements for non-therapeutic indications as judged by the attending physician.
* Regular smoking of more than 5 cigarettes daily use of nicotine-containing products beginning 3 months before study medication administration through the final evaluation.
* If female, the subject is lactating or has a positive pregnancy test at screening and prior to each of the treatment periods. Females of child bearing potential must use a medically acceptable method of contraception throughout the entire study period and for one week after the study is completed. Medically acceptable methods of contraception that may be used by the subject and /or her partner are: oral contraceptives, progestin injection or implant, condom with spermacide, diaphragm with spermicide, IUD, vaginal spermicide Suppository, surgical sterilization of their partner(s) or abstinence. Females taking oral contraceptives must have taken them consistently for at least three months prior to receiving study medication.
* Alcohol, grapefruit beverages or foods or caffeine beverages or foods beginning 1 day before each study medication administration through each study confinement period. Such restricted items include coffee, tea, iced tea, coke®, Pepsi®, Mountain Dew®, Chocolate, brownies, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2004-09; Primary Completion 2004-10 (Actual); Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- aaiPharma, Inc, Chapel Hill, North Carolina, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html